CLINICAL TRIAL: NCT04815265
Title: Efficacy and Safety of Remimazolam for Sedation in ICU Patients Undergoing Mechanical Ventilation: a Single Center, Randomized, Controlled, Non-inferiority Trial
Brief Title: Remimazolam for Sedation in ICU Patients Undergoing Mechanical Ventilation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Nankai Hospital (Other)
Responsible Party: Principal Investigator, Jianbo Yu, Department of Anesthesiology and Critical Care Medicine, Tianjin Nankai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NKYY_YWKT_IRB_2020_007_01
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Sedation
Keywords: Sedation; Mechanical Ventilation
MeSH Terms: interventions — remimazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants in the experimental group received remimazolam for sedation
  Interventions: Drug: Remimazolam
- Control group (Active Comparator): participants in the control group received dexmedetomidine for sedation
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Remimazolam — Remimazolam is used for sedation
  Arms: Experimental group
Drug: Dexmedetomidine — Dexmedetomidine is used for sedation
  Arms: Control group

SUMMARY:
Sedation is a component of the care of critically ill patients who are undergoing mechanical ventilation. Dexmedetomidine induces sedation while preserving a degree of arousability among patients in the intensive care unit (ICU), and its use has resulted in a shorter time to extubation, an increased number of days free from coma or delirium, a reduced incidence of agitated delirium, prevention of delirium, and lower mortality than other agents administered in certain populations. Hypotension and bradycardia are common side effects, which is lethal for the patients with persistent or severe hemodynamic instability.

The pharmacological properties of rimazolom suggest that it is an ideal sedative drug for critically ill patients, but there is no relevant clinical research to confirm it. Therefore, this study mainly discusses the efficacy and safety of remidazolam in ICU patients with mechanical ventilation, so as to provide theoretical basis for individualized sedation treatment of patients with mechanical ventilation.

DETAILED DESCRIPTION:
1. Title: Efficacy and Safety of Remimazolam for Sedation in ICU Patients Undergoing Mechanical Ventilation
2. Research center: Single Center
3. The Design of the study: Randomized, Controlled, Non-inferiority Trial
4. The population of the study: The main inclusion criteria are 18 years old or above, invasive mechanical ventilation is required, and the clinical need is mild to moderate Sedated (RASS score 0 to -3) patients
5. Sample size: Enroll 488 patients (244patients in each group)
6. Interventions: Participants in the test group received remimazolam for sedation, while participants in the control group received dexmedetomidine, The analgesia drug in two group is fentanyl.
7. The aim of the research: To investigate the efficacy and safety of remimazolam for sedation in ICU patients undergoing mechanical ventilation
8. Outcome# 1) Primary outcome# the ratio of the time to reach the target sedation (RASS score, 0 to -3)in the total duration of drug infusion, and the duration of mechanical ventilation. 2)Secondary outcome#; Length of stay in ICU and Length of stay in hospital; Incidence of complications (including re-hospitalization); Total expenses during hospitalization
9. The estimated duration of the study#2-3years

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria are 18 years old or above, invasive mechanical ventilation is required, and the clinical need is mild to moderate Sedated (RASS score 0 to -3) patients.

Exclusion Criteria:

1. Refuse to participate in this study
2. Patients with severe bradycardia (HR<50 bpm)
3. Patients who is pregnancy
4. Patients with brain injury or neurosurgery
5. Patients receiving sedation for treatment indications (such as epilepsy), not to tolerate a ventilator.
6. Patients receiving any study medication within 30 days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to reach targeted sedation goals | an average of 1-2 year
  the ratio of the time to reach the target sedation (RASS score, 0 to -3) in the total duration of drug infusion
the duration of mechanical ventilation | average of 1-2 year
  Duration of mechanical ventilation in ICU

SECONDARY OUTCOMES:
Length of stay in hospital | 2 years
  Length of stay in hospital
Length of stay in ICU | about 2 years
  Length of stay in hospital
Total expenses during hospitalization | 24 months
  Total expenses during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Yu, Study Chair — Tianjin Nankai Hospital

REFERENCES:
- [Background] Shehabi Y, Chan L, Kadiman S, Alias A, Ismail WN, Tan MA, Khoo TM, Ali SB, Saman MA, Shaltut A, Tan CC, Yong CY, Bailey M; Sedation Practice in Intensive Care Evaluation (SPICE) Study Group investigators. Sedation depth and long-term mortality in mechanically ventilated critically ill adults: a prospective longitudinal multicentre cohort study. Intensive Care Med. 2013 May;39(5):910-8. doi: 10.1007/s00134-013-2830-2. Epub 2013 Jan 24. PMID 23344834
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Result] Shehabi Y, Howe BD, Bellomo R, Arabi YM, Bailey M, Bass FE, Bin Kadiman S, McArthur CJ, Murray L, Reade MC, Seppelt IM, Takala J, Wise MP, Webb SA; ANZICS Clinical Trials Group and the SPICE III Investigators. Early Sedation with Dexmedetomidine in Critically Ill Patients. N Engl J Med. 2019 Jun 27;380(26):2506-2517. doi: 10.1056/NEJMoa1904710. Epub 2019 May 19. PMID 31112380
- [Result] Antonik LJ, Goldwater DR, Kilpatrick GJ, Tilbrook GS, Borkett KM. A placebo- and midazolam-controlled phase I single ascending-dose study evaluating the safety, pharmacokinetics, and pharmacodynamics of remimazolam (CNS 7056): Part I. Safety, efficacy, and basic pharmacokinetics. Anesth Analg. 2012 Aug;115(2):274-83. doi: 10.1213/ANE.0b013e31823f0c28. Epub 2011 Dec 20. PMID 22190555